CLINICAL TRIAL: NCT03625167
Title: An Exploratory Randomized Controlled Study to Evaluate the Effect of a Basic Skin Care Product on the Structural Strength of the Dermo-epidermal Junction
Brief Title: Effect of a Basic Skin Care Product on the Structural Strength of the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Jan Kottner (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jan Kottner, Director of the Institute of Clinical Nursing Science, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRC-SP-A31
Record Dates: First submitted 2018-08-01; First posted 2018-08-10 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy Skin
Keywords: skin ageing; suction blister; dermo-epidermal junction
MeSH Terms: interventions — Therapeutics; Petrolatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with petrolatum (Experimental): In each healthy volunteer, one of the two forearms is randomly assigned to the intervention. This forearm is treated with petrolatum for 4 respectively 8 weeks.
  Interventions: Other: Treatment with petrolatum
- Control (No Intervention): The control forearm will remain untreated throughout the study.

INTERVENTIONS:
Other: Treatment with petrolatum — Petrolatum is applied twice daily to the intervention arm.
  Arms: Treatment with petrolatum

SUMMARY:
The main aim of this study is to investigate in a suction blister model, whether the use of a basic skin care formulation increases the mechanical integrity/adhesion of the dermo-epidermal junction.

DETAILED DESCRIPTION:
The process of aging involves numerous structural and functional changes also affecting the skin. The skin fulfills a variety of protective and regulatory functions. Compared to other organs, the skin is constantly exposed to harmful environmental influences. Besides intrinsic factors these external factors may accelerate skin aging. Due to its ageing-related loss of functional capacity the skin becomes susceptible to develop adverse skin conditions and dermatological diseases (e.g. skin dryness, fungal infections). Especially old aged, care depended, and severely ill individuals are at high risk for developing severe skin injuries and wounds (e.g. decubitus, skin tears) with high social and economic impact. Empirical evidence indicates that the reduced adhesion of the dermal-epidermal junction is a major pathophysiological predictor for these types of injuries.

The suction blister model is an artificial and controlled technique for dermal-epidermal separation along the dermo-epidermal junction (DEJ). Empirical evidence suggests that the time of the dermal-epidermal separation (blistering time) is a measure of the dermo-epidermal adhesion. It has been proposed that the blistering time might be a clinically relevant parameter reflecting the mechanical integrity/stability of the dermo-epidermal junction.

Clinical practice guidelines recommend the use of topical skin care products to reduce the risk for pressure ulcer and skin tear development. However, the underlying working mechanisms of most basic skin care products are poorly understood. It is known that topically applied skin care products exhibit physical and chemical effects on and in the uppermost skin layers (e.g. the stratum corneum). Despite a few well known active ingredients (e.g. retinoids, vitamin C) exhibiting effects in the dermis, a particular skin protective effect of the vast majority of daily basic skin care applications on these deeper skin layers is unknown. The primary objective of this study is to test, whether the use of a basic skin care formulation increases the mechanical integrity/adhesion of the dermo-epidermal junction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and/or with stable chronic condition (e.g. controlled hypertension)
* Female,
* 65 to 85 years,
* Caucasian,
* Phototype I to III according to the Fitzpatrick classification,
* Body Mass Index between 20 and 28 kg/m2,
* Non-smoker of at least one year,
* Absence of skin diseases or scars in the skin area of interest,
* Absence of tattoos in the skin area of interest,
* Able to give written informed consent,
* Willing and able to fulfill the study requirements

Exclusion Criteria:

* Known or suspected defect of healing,
* Diabetes mellitus
* Any acute or chronic pathology that may interfere with the trial conduct, from investigator point of view,
* Acute or chronic wounds in the skin area of interest,
* Any skin affection which may interfere with the trial assessment, like urticaria,, psoriasis or scar on investigational areas,
* Medical history of skin cancer,
* History or establishment of diabetes or pre-diabetes,
* Any hyper-sensibility to one of the compounds of the investigational product,
* Any regular treatment which may affect the blood coagulation and hemostasis (anticoagulant medications, NSAID, etc.) before the suction blister induction (Visit 3 and Visit 5), one NSAID to treat headache within four days is allowed
* Any physical treatment (like laser or surgery) on the arms within the last 6 months,
* Use of topical or systemic treatment on the investigational areas within the past 4 weeks (topical hyaluronan, anti-inflammatory drugs, corticoids, retinoids, vitamin C, etc.) that would interfere with assessment and/or investigational treatments,
* Allergy to band-aid or to metals (such as nickel),
* UV sessions or strong sun exposure of the arms during the study period,
* Subject who cannot be contacted easily in case of necessity,
* Current participation in any other clinical study

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kottner, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Clinical Research Center for Hair and Skin Science, Department of Dermatology and Allergy, Charite University Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El Genedy-Kalyoncu M, Richter C, Surber C, Blume-Peytavi U, Kottner J. The effect of a basic skin care product on the structural strength of the dermo-epidermal junction: An exploratory, randomised, controlled split-body trial. Int Wound J. 2022 Feb;19(2):426-435. doi: 10.1111/iwj.13643. Epub 2021 Jun 13. PMID 34121334

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Forearms
Groups:
- Split-Body-Design on Both Forearms. Intervention: Treatment With Petrolatum; Control: No Treatment: In each healthy volunteer, one of the two forearms is randomly assigned to the intervention. This forearm is treated with petrolatum for 4 respectively 8 weeks.
  Treatment with petrolatum: Petrolatum is applied twice daily to the intervention arm.
Period: Overall Study
Arm/Group | Split-Body-Design on Both Forearms. Intervention: Treatment With Petrolatum; Control: No Treatment
Started | 17; 34 Forearms
Completed | 12; 24 Forearms
Not Completed | 5; 10 Forearms
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Units Other Than Participants: Volar forearm
Groups:
- Split-Body-Design on Both Forearms. Intervention: Treatment With Petrolatum; Control: No Treatment: In each healthy volunteer, one of the two forearms is randomly assigned to the intervention. This forearm is treated with petrolatum for 4 respectively 8 weeks.
Arm/Group | Split-Body-Design on Both Forearms. Intervention: Treatment With Petrolatum; Control: No Treatment
Number analyzed (Participants) | 12
Number analyzed (Volar forearm) | 24
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 70.3 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.0 (2.2)
Skin phototype (Fitzpatrick scale) [Count of Participants; unit: Participants] — Skin phototype of participants was classified according the Fitzpatrick classification ranging from phototype I to VI.
  Fitzpatrick Type:
  I: Always burns, never tans (pale skin); II: Usually burns, minimal tanning; III: Occasionally burns, usually tans uniformly; IV: Rarely burns, always tans well; V: Very rarely burns, tans very easily; VI: Never burns, always tans (dark brown/black skin)
  Participants
    Type II | 3
    Type III | 9
Body temperature [Mean (Standard Deviation); unit: degree Celsius] | 36.3 (0.2)
Blood pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 127 (16)
  Diastolic | 83 (9)

OUTCOME MEASURES:

1. Primary Outcome: Blistering Time (Full Blister)
Description: Duration from the start of suction pressure to the development of a full blister (measured in minutes)
Time Frame: Day 28±2, Day 56±2
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Volar forearm
Groups:
- Intervention: Treatment With Petrolatum: Petrolatum was applied twice daily to the randomized volar forearm
- Control: No Treatment: The control forearm remained untreated throughout the study
Arm/Group | Intervention: Treatment With Petrolatum | Control: No Treatment
Number analyzed (Participants) | 12 | 12
Number analyzed (Volar forearm) | 12 | 12
Minutes
  Blistering Time (Full Blister) Day 28±2 | 63 [53 to 94] | 54 [45 to 71]
  Blistering Time (Full Blister) Day 56±2 | 65 [49 to 75] | 62 [42 to 73]

2. Primary Outcome: Blistering Time (First Vesicles)
Description: Duration from the start of suction pressure to the development of first macroscopically visible vesicles (measured in minutes)
Time Frame: Day 28±2, Day 56±2
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Volar forearm
Arm/Group | Intervention: Treatment With Petrolatum | Control: No Treatment
Number analyzed (Participants) | 12 | 12
Number analyzed (Volar forearm) | 12 | 12
Minutes
  Blistering Time (First Vesicles) Day 28±2 | 43 [29 to 69] | 39 [25 to 76]
  Blistering Time (First Vesicles) Day 56±2 | 47 [32 to 69] | 27 [24 to 60]

3. Secondary Outcome: Epidermal Thickness
Description: Optical coherence tomography (OCT) will be used to quantitatively measure changes of the epidermal thickness on the volar forearm
Time Frame: Baseline, Day 28±2, Day 56±2
Measure: Median (Inter-Quartile Range); unit: micrometres (μm)
Units Other Than Participants: Volar forearm
Arm/Group | Intervention: Treatment With Petrolatum | Control: No Treatment
Number analyzed (Participants) | 12 | 12
Number analyzed (Volar forearm) | 12 | 12
micrometres (μm)
  Epidermal Thickness (Baseline) | 78 [65 to 86] | 68 [63 to 80]
  Epidermal Thickness (Day 28±2) | 68 [60 to 84] | 72 [63 to 79]
  Epidermal Thickness (Day 56±2) | 75 [62 to 79] | 71 [65 to 77]

4. Secondary Outcome: Epidermal Hydratation: Stratum Corneum Hydration
Description: Stratum corneum hydration (SCH) was measured with Corneometer® CM 825 (Courage & Khazaka electronic GmbH, Cologne, Germany) and expressed in arbitrary units (AU) (range 0-120 AU) on the volar forearm. Lower values represent reduced skin hydration in the upper skin layer.
Time Frame: Baseline, Day 14±1, Day 28±2, Day 42±2, Day 56±2
Measure: Median (Inter-Quartile Range); unit: Arbitrary Units
Units Other Than Participants: Volar forearm
Arm/Group | Intervention: Treatment With Petrolatum | Control: No Treatment
Number analyzed (Participants) | 12 | 12
Number analyzed (Volar forearm) | 12 | 12
Arbitrary Units
  Stratum corneum hydration (AU) Baseline | 43 [35 to 49] | 40 [35 to 47]
  Stratum corneum hydration (AU) Day 14±1 | 41 [40 to 46] | 36 [34 to 40]
  Stratum corneum hydration (AU) Day 28±2 | 39 [36 to 44] | 36 [33 to 39]
  Stratum corneum hydration (AU) Day 42±2 | 38 [35 to 43] | 36 [33 to 37]
  Stratum corneum hydration (AU) Day 56±2 | 41 [33 to 48] | 35 [32 to 41]

5. Secondary Outcome: Epidermal Hydratation: Epidermal Moisture
Description: Epidermal Moisture (measurement depth 0,5mm) was measured using MoistureMeterEpiD (Delfin Technologies Ltd.). The values are expressed in percentage of local tissue water (0 to 100 %).
Time Frame: Baseline, Day 14±1, Day 28±2, Day 42±2, Day 56±2
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water
Units Other Than Participants: Volar forearm
Arm/Group | Intervention: Treatment With Petrolatum | Control: No Treatment
Number analyzed (Participants) | 12 | 12
Number analyzed (Volar forearm) | 12 | 12
percentage of tissue water
  Epidermal Moisture (%) Baseline | 47 [39 to 54] | 46 [38 to 54]
  Epidermal Moisture (%) Day 14±1 | 46 [42 to 48] | 41 [37 to 46]
  Epidermal Moisture (%) Day 28±2 | 43 [42 to 49] | 41 [38 to 48]
  Epidermal Moisture (%) Day 42±2 | 46 [42 to 58] | 42 [38 to 50]
  Epidermal Moisture (%) Day 56±2 | 47 [42 to 50] | 42 [40 to 43]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant throughout their time of participation (up to 8 weeks). No Adverse Events occurred during the trial.
Description: No Adverse Events occurred during the trial
Groups:
- Intervention: Treatment With Petrolatum: In each healthy volunteer, one of the two forearms is randomly assigned to the intervention. This forearm is treated with petrolatum for 4 respectively 8 weeks. Petrolatum is applied twice daily to the intervention arm.
- Control: No Treatment: The control forearm will remain untreated throughout the study.
Arm/Group | Intervention: Treatment With Petrolatum | Control: No Treatment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT03625167/Prot_SAP_000.pdf